CLINICAL TRIAL: NCT00692068
Title: Relations Between Residual Renal Function and Oxidative and Carbonyl Stress in Peritoneal Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Iwata City Hospital (Other)
Collaborators: University of Shizuoka (Other); Hamamatsu University (Other)
Other Study IDs: ICHKC-2008-1
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Renal Failure
Keywords: residual renal function; oxidative stress; carbonyl stress; peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- A: with residual renal function
- B: without residual renal function

SUMMARY:
Residual renal function is reported to contribute to the survival and cardiovascular disease of peritoneal dialysis patients. Oxidative and carbonyl stress are increased in peritoneal dialysis patients and are associated with cardiovascular risk. The aim of this study was to determine the relations between residual renal function and oxidative and carbonyl stress in peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal failure on peritoneal dialysis

Exclusion Criteria:

* malignancy, peritonitis

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: single dialysis center
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Ryuichi Furuya, M.D., Study Chair — Iwata City Hospital
Locations (1):
- Iwata City Hospital, Iwata, Shizuoka, Japan